CLINICAL TRIAL: NCT02477293
Title: The Efficacy and Safety of Hyeonggaeyeongyo-tang for Chronic Rhinitis According to Pattern Identification in Korean Medicine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Minhee Kim, KMD, Kyung Hee University Hospital at Gangdong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B120014
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Respiratory Tract Diseases; Nose Diseases; Rhinitis
Keywords: Hyeonggaeyeongyo-tang; Chronic rhinitis; Pattern identification; Korean medicine
MeSH Terms: conditions — Respiratory Tract Diseases; Nose Diseases; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyeonggaeyeongyo-tang (Experimental)
  Interventions: Drug: Hyeonggaeyeongyo-tang

INTERVENTIONS:
Drug: Hyeonggaeyeongyo-tang
  Other Names: Hyenggaelong Granule

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Hyeonggaeyeongyo-Tang for chronic rhinitis according to pattern identification in Korean medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed by moderate level of chronic rhinitis for more than 8 weeks

   * At least one of the following conditions: Nasal congestion, rhinorrhea, sneeze, pruritus
   * At least one of the following Moderate abnormality conditions: sleep disturbance; daily activity, physical exercise, leisure activity limitations; work/school work limitations; discomfort with several symptoms
2. Age between 19 and 65 years
3. Able to dialogue
4. Agree with informed consent

Exclusion Criteria:

1. Patients who are taken one of the following drugs for treating rhinitis or acute upper respiratory infections etc

   * Drugs which determined to have negative effect on symptoms of rhinitis or skin prick test (oral or nasal)

     * Short acting anti-histamines / H1 blockers (drug use within lase 1 week)

       * Long acting anti-histamines / H1 blockers (drug use within lase 2 week)

         * Corticosteroids (drug use within lase 1 month) ④ Anti-cholinergic drug (drug use within lase 1 week)

           * Anti-leukotriene drug (drug use within lase 1 week)

             * Decongestants (drug use within lase 1 week) ⑦ Tricyclic antidepressants, phenothiazines (drug use within lase 2 week) ⑧ Non-steroidal analgesics (drug use within lase 1 week) ⑨ Drugs that is judged to be inappropriate for the trial by the researchers
2. Used Korean medicine for treating rhinitis within last 7 days
3. Patients who has severe disease, such as malignant tumor, severe dyslipidemia, liver or kidney dysfunction, anemia, active pulmonary tuberculosis, infection or systemic disease etc
4. Presence of internal nasal obstruction or nasal deformities or history of nasal surgery within 2 months
5. History of active respiratory disease(ex. asthma)
6. Hypertension or Diabetes
7. Experienced immunotherapy or systemic steroid treatments within last 3 months
8. Experienced drug allergic reactions
9. Experienced anaphylactic reactions, during allergen test
10. Female patients who are pregnant or lactating or have the chances of pregnancy
11. Patients who are participated other clinical trials within last 1 month
12. Patients who are unable to participate the trial (paralysis, severe mental or psychological illness, dementia, drug addiction, unable to make to participate in the trial, severe visual or auditory dysfunction, unable to visit hospital regularly, unable to communicate through spoken or written Korean etc)
13. Patients who are judged to be inappropriate for the clinical study by the researchers

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 'Total nasal symptom score (TNSS)' | At baseline, Day 2(Scheduled within a week of baseline), Week 3, 5, 9, 13
Change from baseline in 'pre KiFDA-AR ver 2.0' Questionnaire | At baseline, Day 2(Scheduled within a week of baseline), Week 3, 5, 9, 13

SECONDARY OUTCOMES:
Pattern Diagnosis by 'Cold-heat Pattern Identification Questionnaire' | Day 2(Scheduled within a week of baseline)
  Pattern Diagnosis(either cold or heat pattern) based on the results of Cold-heat Pattern Identification Questionnaire
Change from baseline in 'Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)' | At baseline, Day 2(Scheduled within a week of baseline), Week 3, 5, 9, 13
Pattern diagnosis by doctor of Korean medicine by traditional Korean medicine doctor's four examination | Day 2(Scheduled within a week of baseline)
  Pattern Diagnosis(either wind-heat or wind-cold pattern) based on the results of traditional Korean medicine doctor's four examination(questioning/history taking, inspection, auscultation (listening) & olfaction (smelling), and palpation)
Diagnosis of secondary complications of chronic rhinitis (allergic rhinitis) by skin prick test | Day 2(Scheduled within a week of baseline)
  Observed the allergic reaction for assessing the allergenicity of patients with allergic rhinitis
Change from baseline in total immunoglobulin E (IgE) | Day 2(Scheduled within a week of baseline), Week 5
Change from baseline in 'Heart Rate Variability' | Day 2(Scheduled within a week of baseline), Week 5
Change from Baseline in 'Ryodoraku values' | Day 2(Scheduled within a week of baseline), Week 5
  Investigate the different changes on autonomic nervous system from Ryodoraku value. The 12 measured Ryodoraku points are 6 on the hand(represented as H) and 6 on the feet(represented as F).
Diagnosis of secondary complications of chronic rhinitis (allergic rhinitis and rhino-sinusitis) by Waters, Caldwell, and lateral view (paranasal sinus 3P) | Day 2(Scheduled within a week of baseline)
Change from baseline in 'Perceived Stress Scale' | Day 2(Scheduled within a week of baseline), Week 5
Change from baseline in eosinophil count level | Day 2(Scheduled within a week of baseline), Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Kyu Ko, KMD, PhD, Study Chair — Kyunghee University
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Kim MH, Son J, Nam HJ, Ko SG, Choi I. Hyeonggaeyeongyo-Tang for Treatment of Allergic and Nonallergic Rhinitis: A Prospective, Nonrandomized, Pre-Post Study. Evid Based Complement Alternat Med. 2016;2016:9202675. doi: 10.1155/2016/9202675. Epub 2016 Sep 6. PMID 27698676